CLINICAL TRIAL: NCT06927128
Title: Single - Center Phase II Clinical Study: Efficacy Evaluation of Neoadjuvant Chemotherapy With Gemcitabine and Cisplatin in High - Risk Upper Tract Urothelial Carcinoma
Brief Title: Neoadjuvant Chemotherapy in High - Risk Upper Tract Urothelial Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-NAC-UTUC
Record Dates: First submitted 2025-03-16; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: UTUC; NAC
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Gemcitabine Plus Cisplatin Chemotherapy Group (Experimental): Participants receive intravenous gemcitabine (1000 mg/m²) on days 1 and 8, followed by intravenous cisplatin (70 mg/m²) on day 1, every 3 weeks for 4 cycles. This neoadjuvant chemotherapy is administered prior to planned radical nephroureterectomy.
  Interventions: Drug: Gemcitabine, Cisplatin

INTERVENTIONS:
Drug: Gemcitabine, Cisplatin — Gemcitabine (1000mg/m²) and cisplatin (70mg/m²). Gemcitabine is used on the 1st and 8th days of a 21 - day cycle, and cisplatin is used on the 2nd day of the cycle. A total of 3 - 4 cycles are carried out.A dose reduction to 60% of the original dose (adjusted to 0.6 times the initial dose) will be implemented if deemed clinically necessary, contingent upon meeting either of the following criteria: 1) occurrence of grade 3 or higher treatment-related adverse events as per CTCAE v5.0 guidelines, or 2) evidence of renal impairment manifested by a ≥40% decline in glomerular filtration rate (GFR) from baseline measurements.

SUMMARY:
Upper urinary tract urothelial carcinoma (UTUC) represents a rare yet aggressive malignancy associated with a dismal prognosis. At the point of diagnosis, nearly half of the patients already have invasive disease, and over 70% present with high-grade UTUC. Currently, radical nephroureterectomy (RNU) remains the gold standard of care for high-risk UTUC.

Previous investigations have demonstrated that, in contrast to RNU alone, chemotherapy can effectively reduce the disease recurrence rate and mortality. Moreover, it may confer benefits to patients' overall survival (OS) without impeding the implementation of subsequent definitive surgical treatment. However, the majority of these studies are predominantly retrospective analyses. Although they can, to some degree, reflect the clinical value of neoadjuvant chemotherapy, due to inherent limitations in study design and other confounding factors, there is still a paucity of prospective research evidence for further validation.

Considering that RNU can cause a decline in renal function in patients, and in light of prospective trial outcomes, preoperative neoadjuvant chemotherapy (NAC) has emerged as a preferred treatment option for chemotherapy-eligible UTUC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high - risk upper tract urothelial carcinoma (UTUC). For mixed - type tumors, the histological type should be mainly urothelial carcinoma (≥50%), or urine cytology is positive and imaging diagnosis supports UC.
* Clinically non - metastatic urothelial carcinoma (N≤1 M0), determined by imaging examinations (CT or MRI) of the chest/abdomen/pelvis.
* Patients must plan to undergo radical nephroureterectomy (RNU).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Patients are potential beneficiaries of cisplatin - based neoadjuvant chemotherapy, with relatively good renal function (GFR≥45ml/min) and able to tolerate drug treatment and surgery.
* Sufficient organ and bone marrow function determined by screening tests.
* Recovered from any reversible toxicity of previous surgery.
* At least 18 years old on the date of registration.
* Informed of the study nature and signed the informed consent form.

Exclusion Criteria:

* Imaging - identified ≥N2 disease or metastatic disease (M1).
* History of invasive or lymph node - positive or metastatic urothelial carcinoma or invasive contralateral upper tract carcinoma within 2 years before registration.
* Patients with only one kidney, or cisplatin intolerant patients.
* Participating in other interventional clinical trials at the time of registration.
* History of non - urothelial malignancies, except those who have been disease - free for at least 1 year as judged by the treating oncologist. History of adequately treated (at the discretion of the treating oncologist) basal cell or squamous cell skin cancer or in - situ cervical cancer is allowed.
* Pregnant or lactating women. Reproductive - potential women/men must agree to use effective contraception methods.
* Any other medical conditions that make the treating doctor consider their participation in the study inappropriate.

Withdrawal/Termination Criteria

* Investigator - determined Withdrawal:
* Tumor recurrence or progression during the clinical trial, and the investigator determines that the subject needs new treatment (such as immediate tumor resection or systemic anti - tumor treatment) and is not suitable to continue the trial. If the investigator judges that the subject can still receive treatment or follow - up for efficacy after tumor recurrence, the subject may not be withdrawn for the time being.
* The subject develops comorbidities, complications, or special physiological changes that are not suitable for continuing the trial.
* Poor compliance of the subject affecting safety and efficacy evaluation:
* The subject does not take medicine or undergo examinations as required.
* The subject uses other drugs or foods that affect safety evaluation.
* The subject has other behaviors that affect the test results.
* Unbearable toxicity, other adverse events, or serious adverse events occur, and the subject is not suitable to continue the trial.
* A grade 3 adverse event related to the study drug occurs and persists for more than 12 days after taking sufficient treatment measures.
* Systemic metastasis or progression is detected during the drug - administration observation period or the surgical period.
* Subject - initiated Withdrawal: Subjects have the right to withdraw from the trial midway according to the informed consent form. If the subject does not withdraw the informed consent but no longer accepts trial drug administration and examinations or is lost to follow - up, it is also regarded as withdrawal. All withdrawn subjects should try to complete the corresponding observation content of the last visit as specified in the protocol. The reason for termination should be noted in the original document. If the subject withdraws due to an adverse event, appropriate treatment should be provided and recorded in the original record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate（pRR） | At the time of pathological report issuance，approximately within 7-10 business days after surgery
  defined as postoperative pathology <ypT2N0

SECONDARY OUTCOMES:
Pathological complete response rate (pCR) | At the time of pathological report issuance，approximately within 7-10 business days after surgery
  defined as postoperative pathology <ypT1N0
Imaging response rate | From the date of the first chemotherapy administration until 2 weeks after the last chemotherapy session, assessed up to 11-14 weeks.
  defined as tumor size reduction observed on imaging comparisons between pre- and post-chemotherapy assessments, with any decrease classified as a positive response.Tumor size reduction, measured as the change in the longest diameter of the primary tumor via computed tomography (CT) scan according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.
Surgery completion rate | From chemotherapy initiation to surgical resection.Patients should undergo definitive surgery within 6 weeks ( ± 2 weeks) following completion of neoadjuvant chemotherapy
  Proportion of patients undergoing surgery
Overall survival (OS) | From the date of surgery until the date of death or loss to follow-up, with a maximum follow-up period of 2 years.
  defined as the duration from the date of surgical resection to the occurrence of death from any cause
Cancer - specific survival (CSS) | From the date of diagnosis until the date of death from urothelial carcinoma or last documented follow-up, with a maximum follow-up period of 2 years.
  defined as the time from diagnosis to death directly attributable to the primary cancer or its metastases, excluding mortality from unrelated causes
Recurrence - free survival (RFS) | From the date of surgical resection until the date of disease recurrence (radiographically or pathologically confirmed) or death from any cause, whichever occurs first, with a maximum follow-up of 2 years.
  defined as the time from post-surgery to the first documented evidence of local/regional recurrence, distant metastasis, or death from any cause, whichever occurs first

OTHER OUTCOMES:
the efficacy by detecting the chromosomal instability (CIN) of blood and urine exfoliated cell DNA | From the time of collecting the first blood and urine specimens until the time of collecting blood and urine specimens before surgery, assessed up to 15-18 weeks.
  Predicting the efficacy by detecting the chromosomal instability (CIN) of blood and urine exfoliated cell DNA

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided